CLINICAL TRIAL: NCT05071573
Title: Optimised Electronic Patient Records to Improve Clinical Monitoring of HIV-positive Patients in Rural South Africa (MONART Trial)
Brief Title: Optimised Electronic Patient Records to Improve Clinical Monitoring of HIV-positive Patients in Rural South Africa
Acronym: MONART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sussex (Other)
Collaborators: Africa Health Research Institute (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ER/BSMS9B5G/4
Record Dates: First submitted 2021-09-15; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections
Keywords: HIV; HIV viral load; HIV drug resistance; Treatment failure; Virological suppression
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: An innovative effectiveness-implementation hybrid cluster-randomised trial in 10 clinics to evaluate the effectiveness of the interventions for improving VLM and virological suppression compared with current care. Clinics will be randomly allocated to either the intervention (Quality improvement package, viral load champion, and augmentation of TIER.Net) or current care.
Masking Description: The 10 clinics will be randomly allocated to the intervention (5 clinics) and control (5 clinics) arms. Randomisation will be stratified on clinic size, defined by the number of HIV-related visits per month (2 strata). Restricted randomisation will be used to ensure balance between study arms on the following important covariates: proportion of HIV patients who are male; proportion of HIV patients who are aged <25 years. A computer programme will be used to prepare a list of all permissible randomised combinations; community leaders will be invited to make a random selection from the list at a public ceremony. The randomisation list will be prepared by an independent statistician and will be concealed until after randomisation. It will not be possible to blind the research staff and nurses to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Quality improvement package Identification of a viral load champion whose role will include tracing and recalling patients who need further assessments of their VL or switch to second-line regimen.
  QIP to address process and clinic impediments to VLM as well as training in antiretroviral treatment monitoring guidelines Training in the use of enhanced TIER.Net technology developed as part of the trial and how to access reports on the dashboard system.
  Augmentation of TIER.Net with a dashboard system VL results will be imported into TIER.Net daily from the National Health Laboratory Service which will be linked to patients in TIER.Net based on multiple exclusive and linked deterministic rules using a combination of variables such as name, surname, sex, date of birth, date of visit, NHLS lab number, facility and folder number. The information contained in TIER.Net will be used to develop a dashboard which summarises viral load data at individual and clinic level.
  Interventions: Other: Optimised electronic patient records
- Control arm (No Intervention): Viral load results are manually captured on to the TIER.Net system with filing of the paper results in patients' clinical notes for nurses' review during routine appointments. This is used to produce a monthly enrolment and quarterly cohort reports for the central monitoring of the ART programme.

INTERVENTIONS:
Other: Optimised electronic patient records — Viral load champions trained in the monitoring of patient on antiretroviral therapy to aid prompt identification of virological failure and institution of appropriate clinical management
  Arms: Intervention arm

SUMMARY:
In our formative research, analysis of antiretroviral treatment (ART) data manually entered in the Three Interlinked Electronic Registers (TIER.Net) showed poor viral load monitoring (VLM) and inadequate management of virological failure in HIV-positive patients on ART in rural KwaZulu-Natal, South Africa. ART interruption was high, with nearly half of patients falling out of care within 5 years of starting ART. Non-Nucleoside reverse transcriptase pre-treatment drug resistance exceeds 10% in the setting; the threshold required to trigger in a change in first-line ART using the public health approach. These factors are contributory to increasing HIV drug resistance (HIVDR) in this setting. HIVDR is associated with increased morbidity and mortality with the risk of transmitting drug-resistant HIV to sexual partners. The investigators presented these findings to healthcare providers, policy makers and community representatives with brainstorming of health system challenges and potential interventions. This study aims to complement these findings by investigating the clinical and process impediments in VLM within the health system and to develop a quality improvement package (QIP) to address the gaps. The stakeholders recommended such QIP would utilise the viral load (VL) champion model, a named healthcare provider who would be the focal point for ensuring proper administrative management of viral load tests and results through identification of those who need tests and triaging of results for action. This QIP will be supported by technological enhancement of the routine clinic-based TIER.Net software which will allow daily automatic import of results from the National Health Service Laboratory (NHLS) to TIER.Net and development of a dashboard system to support VLM. In addition, results of contact tracing will be recorded and followed up pro-actively if not initially successful.

The investigators will evaluate the effectiveness of these interventions compared to standard care for improving VLM and virological suppression using an innovative effectiveness-implementation hybrid cluster-randomised design in 10 clinics. A within-trial health economics analysis will be undertaken using recommended methods to examine the cost-effectiveness of the intervention compared to standard care.

DETAILED DESCRIPTION:
South Africa has the biggest HIV treatment programme in the world with 7.7 million individuals living with HIV and 62% currently receiving ART within a stretched health system. VLM has been part of the public ART programme since roll-out in 2004 and requires people with HIV initiating ART to have a VL measured at 6 months and 12 months after ART initiation and 12-monthly thereafter if virologically suppressed. Those with a VL ≥ 1000 HIV-1 RNA copies/mL should be retested after 3 months of adherence counselling support, and then either retained on first-line therapy if re-suppressed or switched to second-line therapy if VL ≥ 1000 copies/mL.

However, little is known about how these VL guidelines are being used in clinical decision-making in public ART programmes in sub-Saharan Africa. In formative research utilising an electronic database, the Three Interlinked Electronic Register (TIER.Net), of a programmatic ART cohort in rural KwaZulu-Natal, the investigators observed infrequent VLM and sub-optimal management of virological failure. The study showed that only 34% of patients had a viral load documented after 12 months on ART. Only 20% of individuals in the cohort were confirmed to have virologic re-suppression or change to second line therapy after virologic failure, and those that did change therapy did so a median of one year after virologic failure. With the expansion in the indications for ART use, such delays are likely to have significant deleterious individual and public health impacts through effects on patient morbidity, accumulation of drug resistance, and persistent risk of HIV transmission in the setting.

The investigators hypothesise that a staff-centred quality improvement package (QIP) and technological augmentation of an existing electronic ART database (TIER.Net) would result in optimal VLM of patients on ART, prompt clinical management of virological failure and an overall improvement in virological suppression.

Main trial objective

The main objective is to evaluate the impact of a combination of interventions that includes a staff-centred quality improvement package, designated viral load monitoring champion, and augmentation of TIER.Net with a dashboard system will lead to improvement in viral load monitoring and virological suppression over a period of 12 months in comparison to the current standard of care.

Secondary objectives

* To identify health system specific gaps in VLM.
* To evaluate the cost and cost effectiveness of the intervention compared to standard care

ELIGIBILITY:
Inclusion Criteria:

* All nursing care staff employed at the health facilities are eligible for inclusion to receive the quality improvement intervention
* Willing to provide informed consent
* Work in one of the ten facilities randomised for the study
* Involved in HIV patient care
* Patients receiving care from participating clinics must be aged 16 years and above to be included in the study

Exclusion Criteria:

* Expecting to relocate or change jobs during the study duration
* Unwilling or unable to provide informed consent/refusal to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of all patients who have a VL measurement and are virally suppressed (composite outcome) after 12 months of follow up. | 12 months
  Viral suppression defined as VL < 50 c/mL

SECONDARY OUTCOMES:
Proportion of all patients with at least one documented VL in TIER.Net during the trial follow up. | 12 months
  Participant has viral load results present in TIER.Net
Proportion with VL ≥50 c/mL during follow up | 12 months
  Participants who did not achieve viral suppression at the end of follow up
Proportion with a repeat test within 3 months amongst patients with VL ≥1000 c/mL | 12 months
  Guidelines recommend repeat VL after 3 months in patients with VL ≥1000 c/mL and if VL is still ≥1000 c/mL, to switch to second-line ART. This outcome assesses adherence to treatment guidelines.
Time from first VL ≥1000 c/mL to repeat VL | 12 months
  Guidelines recommend repeat VL after 3 months in patients with VL ≥1000 c/mL and if VL is still ≥1000 c/mL, to switch to second-line ART. This outcome assesses adherence to treatment guidelines.
Proportion switching to second-line ART after two consecutive VL≥1000 c/mL measured ≤3 months apart | 12 months
  Guidelines recommend repeat VL after 3 months in patients with VL ≥1000 c/mL and if VL is still ≥1000 c/mL, to switch to second-line ART. This outcome assesses adherence to treatment guidelines.
Cost-effectiveness of the intervention | 12 months
  A within-trial health economics analysis will be undertaken using recommended methods to examine the cost-effectiveness of the intervention compared to standard care. The investigators will estimate the cost of the intervention, including implementation of QIP and the augmentation of TIER.net. The investigators will collect cost data on ART, tests, consultations and hospitalisations over the 12-month period. The primary cost-effectiveness analyses will be conducted using the proportions of patients who did not have a VL measurement; patients with VL documented in clinical charts; and patients with VL measurement but no results in clinical charts.

CONTACTS AND LOCATIONS:
Overall Officials: Collins Iwuji, MD, Principal Investigator — University of Sussex
Locations (1):
- Africa Health Research Institute, Mtubatuba, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Iwuji C, Osler M, Mazibuko L, Hounsome N, Ngwenya N, Chimukuche RS, Khoza T, Gareta D, Sunpath H, Boulle A, Herbst K. Optimised electronic patient records to improve clinical monitoring of HIV-positive patients in rural South Africa (MONART trial): study protocol for a cluster-randomised trial. BMC Infect Dis. 2021 Dec 20;21(1):1266. doi: 10.1186/s12879-021-06952-5. PMID 34930182